CLINICAL TRIAL: NCT07088094
Title: The Clinical Study of Bone-patellar Tendon-bone and Quasi-anatomical Meniscus Allograft Transplantation Technique
Acronym: BPTB，Meniscus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Principal Investigator, YujiakuoTHU, Principal Investigator, Beijing Tsinghua Chang Gung Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25076-3-01; 12110000318301495P (Other: Beijing Tsinghua Changgung Hospital)
Record Dates: First submitted 2025-05-18; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Meniscal Tears; ACL - Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bone-patellar tendon-bone allograft transplantation (Experimental): Bone-patellar tendon-bone allograft transplantation
  Interventions: Procedure: bone-patellar tendon-bone or meniscus allograft transplantation techniques
- Control group (No Intervention): non-surgical or conservative treatment group
- Quasi-anatomical meniscus allograft transplantation (Experimental): Quasi-anatomical meniscus allograft transplantation
  Interventions: Procedure: Quasi-anatomical meniscus allograft transplantation

INTERVENTIONS:
Procedure: bone-patellar tendon-bone or meniscus allograft transplantation techniques — This clinical study follows an interventional design, focusing on the evaluation of bone-patellar tendon-bone and quasi-anatomical meniscus allograft transplantation techniques。
  Arms: Bone-patellar tendon-bone allograft transplantation
Procedure: Quasi-anatomical meniscus allograft transplantation — Quasi-anatomical meniscus allograft transplantation
  Arms: Quasi-anatomical meniscus allograft transplantation

SUMMARY:
This clinical study investigates the outcomes of bone-patellar tendon-bone and quasi-anatomical meniscus allograft transplantation techniques in patients requiring joint reconstruction. The study aims to assess the safety, efficacy, and functional improvements following these transplant procedures, utilizing donor tissues to restore joint function and alleviate pain in individuals with severe knee damage. Participants will undergo the transplantation procedure and be monitored for post-operative recovery, complications, and long-term outcomes, including joint stability and mobility. The study seeks to provide valuable insights into the effectiveness of these advanced surgical techniques for knee joint repair.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-50 years
* Clinical diagnosis of symptomatic meniscal deficiency and anterior cruciate ligament injury (complete rupture or severe damage)
* Failure of conservative treatment (e.g., physical therapy, analgesia) for ≥6 months
* Stable knee joint (no ligamentous instability confirmed via clinical exam and MRI)
* Willingness to comply with postoperative rehabilitation and follow-up evaluations

Exclusion Criteria:

* Severe tibiofemoral osteoarthritis (Kellgren-Lawrence grade ≥3)
* History of prior knee infection or septic arthritis
* Inflammatory arthritis (e.g., rheumatoid arthritis, gout)
* BMI ≥35 kg/m²
* Pregnancy or planning pregnancy during the study period
* Concurrent full-thickness chondral defects (Outerbridge grade III-IV) in the affected compartment
* Inability to undergo MRI (e.g., claustrophobia, metallic implants)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative Complications Unit of Measure | 2 years
  Unit of Measure: Percentage of patients with complications (e.g., infection, graft failure, arthrofibrosis)
  Description: This measure evaluates the incidence of postoperative complications in patients undergoing bone-patellar tendon-bone and quasi-anatomical meniscus allograft transplantation techniques. The complications will be classified according to the Clavien-Dindo Classification for surgical complications, with clinical evaluations using physical examination and imaging to assess the occurrence of adverse events. The results will be reported as the percentage of patients experiencing any form of complication during the postoperative period.
  Measurement Tool: Clavien-Dindo Classification for surgical complications, clinical evaluation through physical examination, and imaging studies.
Functional Improvement in Knee Joint Unit of Measure-Knee Society Score (KSS) | 2 years
  Unit of Measure: Improvement in functional scores (0-100 scale)
  Description: This measure evaluates the improvement in knee function following bone-patellar tendon-bone and quasi-anatomical meniscus allograft transplantation techniques. Functional outcomes will be assessed using the Knee Society Score (KSS)
  What it measures:
  Knee Score (0-100): Knee-specific symptoms, alignment, stability. Function Score (0-100): Walking distance, stair-climbing, use of aids. Score Meaning: Higher = Better outcome. Note: Reported as two separate scores (not combined).
  Measurement Tool: Knee Society Score (KSS) and Lysholm Knee Score. The scale use a 0-100 range, where higher scores always indicate better knee function/health.
Functional Improvement in Knee Joint Unit of Measure-Lysholm Knee Score | 2 years
  Unit of Measure: Improvement in functional scores (0-100 scale)
  Description: This measure evaluates the improvement in knee function following bone-patellar tendon-bone and quasi-anatomical meniscus allograft transplantation techniques. Functional outcomes will be assessed using Lysholm Knee Score.
  Full Name: Lysholm Knee Scoring Scale Range: 0-100 What it measures: Stability, pain, daily function. Score Meaning: Higher = Better outcome.
  Measurement Tool: Lysholm Knee Score. The scale use a 0-100 range, where higher scores always indicate better knee function/health.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Jiang D, Ao YF, Gong X, Wang YJ, Luo H, Chen LX, Wang HJ, Xie X, Zhang JY, Yu JK. Double-bundle anterior cruciate ligament reconstruction using bone-patellar tendon-bone allograft: technique and 2- to 5-year follow-up. Am J Sports Med. 2012 May;40(5):1084-92. doi: 10.1177/0363546512440686. Epub 2012 Apr 2. PMID 22472270
- [Result] Wang DY, Lee CA, Zhang B, Li YZ, Meng XY, Jiang D, Yu JK. The immediate meniscal allograft transplantation achieved better chondroprotection and less meniscus degeneration than the conventional delayed transplantation in the long-term. Knee Surg Sports Traumatol Arthrosc. 2022 Nov;30(11):3708-3717. doi: 10.1007/s00167-022-06982-9. Epub 2022 Apr 28. PMID 35484433

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-17): https://cdn.clinicaltrials.gov/large-docs/94/NCT07088094/Prot_SAP_000.pdf
  • Informed Consent Form (2025-03-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT07088094/ICF_001.pdf